CLINICAL TRIAL: NCT00616434
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Avonex® in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: A Phase 2 Study of Interferon Beta-1a (Avonex®) in Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108UC201; 2007-004867-22 (EudraCT Number); NCT00750490 (obsolete NCT alias)
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Active Ulcerative Colitis
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interferon beta-1a (Experimental): Interferon beta-1a 30 µg intramuscular (IM) injection twice weekly for 12 weeks
  Interventions: Drug: BG9418 (Interferon beta-1a)
- Placebo (Placebo Comparator): Placebo IM injection twice weekly for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BG9418 (Interferon beta-1a) — Avonex IM injection, self-administered per protocol
  Other Names: Avonex®
  Arms: Interferon beta-1a
Drug: Placebo — Placebo IM injection, self-administered per protocol.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the clinical activity of interferon beta-1a in participants with moderate to severe ulcerative colitis (UC). Secondary objectives of this study are to determine (i) the safety and tolerability of interferon beta-1a in participants with moderate to severe UC, and (ii) the percentage of participants, with a decrease in the Simple Clinical Colitis Activity Index (SCCAI) score of ≥3 points at Week 8.

ELIGIBILITY:
Key Inclusion Criteria:

* Established diagnosis of ulcerative colitis (UC) for ≥6 months

  * 20 cm active disease at Screening endoscopy
* Must have active UC with a Mayo Score/Disease Activity Index (DAI) of 6 to 13 points and moderate to severe disease on endoscopy (Mayo endoscopic score of at least 2) despite prior or concomitant treatment
* Colonoscopy within past 5 years for extent of disease and to exclude polyps
* For subjects with UC for more than 10 years, colonoscopy with appropriate biopsies within 1 year prior to Screening to exclude dysplasia and neoplasia.
* Must be willing and able to practice effective birth control during the study and for 1 month after the last dose of study treatment.

Key Exclusion Criteria:

* Diagnosis of indeterminate colitis or Crohn's disease
* Need for imminent surgery
* Diagnosis of primary sclerosing cholangitis or toxic megacolon
* Hemoglobin ≤9 g/dL
* White blood cell count < 3500 cells/mm^3
* Lymphocyte count <1000 cells/µL
* Platelet count <100,000 cells/µL
* Female subjects who are pregnant or who wish to become pregnant during the study, or who are lactating
* Known symptomatic colonic stricture
* Stool cultures positive for enteric infection
* History of malignant disease
* History of major abdominal surgery (e.g., gastrectomy) within past 5 years
* History of small bowel or colonic obstruction or resection
* History of drug or alcohol abuse (as defined by the Investigator) within 2 years prior to Screening
* Use of anti-diarrheal agents during the screening period
* Previous participation in this study
* Previous treatment with interferon beta or other interferon products

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (35):
- United States (5):
  - Investigator, Birmingham, Alabama
  - Investigator, Lakewood, Colorado
  - Investigator, Bristol, Connecticut
  - Investigator, Wellesley Hills, Massachusetts
  - Investigator, Oklahoma City, Oklahoma
- Canada (3):
  - Investigator, Calgary, Alberta
  - Investigator, Kelowna, British Columbia
  - Investigator, Winnipeg, Manitoba
- Czechia (6):
  - Investigator, Hradec Králové
  - Investigator, Ostrava
  - Investigator, Parbudice
  - Investigator, Prague
  - Investigator, Slaný
  - Investigator, Teplice
- Hungary (4):
  - Investigator, Budapest
  - Investigator, Eger
  - Investigator, Szeged
  - Investigator, Székesfehérvár
- Poland (6):
  - Investigator, Lublin
  - Investigator, Pruszków
  - Investigator, Sopot
  - Investigator, Torun
  - Investigator, Warsaw
  - Investigator, Wroclaw
- Russia (9):
  - Investigator, Kazan'
  - Investigator, Krasnodar
  - Investigator, Lipetsk
  - Investigator, Moscow
  - Investigator, Nizhny Novgorod
  - Investigator, Rostov-on-Don
  - Investigator, Saint Petersburg
  - Investigator, Saratov
  - Investiator, Yaroslavl
- Slovakia (2):
  - Investigator, Nitra
  - Investigator, Trenčín

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interferon Beta-1a | Placebo
Started | 62 | 61
Completed | 56 | 53
Not Completed | 6 | 8
Not completed — Adverse Event | 5 | 2
Not completed — Physician Decision | 0 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a | Placebo | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Full Range); unit: years] | 41.1 [21 to 64] | 41.0 [20 to 65] | 41.0 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 45
  Male | 43 | 35 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinical Response
Description: Clinical response is defined as a decrease from baseline in the total Mayo score of at least 3 points and at least 30%, accompanied by a decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore of 1 or less. Baseline was defined as the score collected during the screening period. The Mayo Score/Disease Activity Index (DAI) measures disease activity through assessment of 4 items: stool frequency, rectal bleeding, endoscopy findings, and Physician Global Assessment (PGA). Each item of the score is assessed on a 4-point scale, 0, 1, 2, or 3, with a higher score representing greater severity. In this study, the endoscopy subscore was expanded to a 5-point scale to increase sensitivity in this important dimension of the disease (0=normal/inactive disease, 4=deep ulceration). The Total Mayo Score can therefore range from 0 to13 points.
Time Frame: Baseline and Week 8
Population: Intent-to-treat (ITT): Defined as all randomized participants who received at least one dose of study treatment for whom a baseline measure was available.
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta-1a | Placebo
Number analyzed (Participants) | 62 | 61
percentage of participants | 53 | 44

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE, can therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. All AE's were analyzed based on the principle of treatment emergence. An AE was regarded as treatment-emergent if it was not present prior to receiving the first injection but subsequently appeared, or if it was present prior to receiving the first injection and subsequently worsened in severity.
Time Frame: Up to 16 weeks
Population: Safety Population; participants who were randomized and received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Interferon Beta-1a | Placebo
Number analyzed (Participants) | 62 | 61
participants | 52 | 35

3. Secondary Outcome: Percentage of Participants With a Decrease on Simple Clinical Colitis Activity Index (SCCAI) of ≥3 Points at Week 8
Description: The SCCAI measures disease activity as defined by both participants and examiners and includes the following 13 items: general well-being, abdominal pain, bowel frequency, stool consistency, bleeding, anorexia, nausea or vomiting, abdominal tenderness, extra-intestinal complications (eye, mouth, joint, skin), temperature, sigmoidoscopic assessment, nocturnal bowel movements, and urgency of defecation. Scores range from 0 to 19 points, and scores <2.5 have been shown to correlate with Patient-Defined Remission, and a decrease of >1.5 points from Baseline correlates with Patient-Defined Significant Improvement. Baseline is defined as the mean of the screening and visit 1 scores.
Time Frame: Baseline and Week 8
Population: Intent-to-treat (ITT): Defined as all randomized participants who received at least one dose of study treatment for whom a baseline SCCAI ≥ 3 was available.
Measure: Number; unit: percentage of participants
Arm/Group | Interferon Beta-1a | Placebo
Number analyzed (Participants) | 61 | 61
percentage of participants | 64 | 46

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Interferon Beta-1a | Placebo
Serious Adverse Events (participants affected / at risk) | 1/62 | 3/61
Other Adverse Events (participants affected / at risk) | 44/62 | 20/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=62) | Placebo (N=61)
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 2
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=62) | Placebo (N=61)
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 6
Headache (Nervous system disorders) | 11 | 3
Hypertension (Vascular disorders) | 3 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Influenza Like Illness (General disorders) | 25 | 6
Pyrexia (General disorders) | 8 | 2
Malaise (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.